CLINICAL TRIAL: NCT01303913
Title: Composite Analysis on Factors That Predict Oxygen Desaturation During Walking in COPD
Brief Title: Predicting Oxygen Desaturation in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Type: Observational
Sponsor: Villa Pineta Hospital (Other)
Responsible Party: Villa Pineta Hospital, Villa Pineta Hospital
Other Study IDs: VP03-2010
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: COPD
Keywords: COPD; Oxygen desaturation; Walking test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Walking desaturation group: COPD patients that at the end of 6MWT have SO2 nadir <88-90%
- Walking No-desaturation group: COPD patients that at the end of 6MWT have SO2 nadir >88-90%

SUMMARY:
Oxygen desaturation (SO2 < 88-90%) during walking is a common clinical feature of Chronic Obstructive Pulmonary Disease (COPD) patients. By a predicted analysis our study is aimed to evaluate anthropometric and functional characteristics of COPD patients correlated with oxygen desaturation during Six-minute walking test (6MWT).

ELIGIBILITY:
Inclusion Criteria:

* COPD patients
* Ability to perform 6MWT
* Normal oxygen saturation at rest and at the begin of 6MWT

Exclusion Criteria:

* No-COPD patients
* Chronic Respiratory Failure patients in Long-term oxygen therapy (LTOT)
* Any co-morbidities

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-06; Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation nadir (SO2 nadir) | Measured at the end of 6MWT
  Measured by change in percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Crisafulli, MD, PhD, Principal Investigator — Villa Pineta Hospital
Locations (1):
- Villa Pineta Hospital, Pavullo nel Frignano, Modena, Italy

REFERENCES:
- [Derived] Crisafulli E, Iattoni A, Venturelli E, Siscaro G, Beneventi C, Cesario A, Clini EM. Predicting walking-induced oxygen desaturations in COPD patients: a statistical model. Respir Care. 2013 Sep;58(9):1495-503. doi: 10.4187/respcare.02321. Epub 2013 Jan 29. PMID 23362168